CLINICAL TRIAL: NCT02383069
Title: Pulmonary Rehabilitation in Asthmatic Pediatric Patients: Randomized Clinical Trial
Brief Title: Pulmonary Rehabilitation in Asthmatic Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fernanda de Cordoba Lanza (Other)
Collaborators: University of Nove de Julho (Other); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Federal University of Minas Gerais (Other)
Responsible Party: Sponsor-Investigator, Fernanda de Cordoba Lanza, PhD, Professor, University of Nove de Julho
Organization: University of Nove de Julho (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPR-UNI9
Record Dates: First submitted 2015-02-10; First posted 2015-03-09 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Asthmatic; Children
Keywords: Pulmonary rehabilitation; Asthma; Children; Teenager; Physical capacity
MeSH Terms: conditions — Asthma | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will have supervised rehabilitation program held twice a week, each session will have 60 minutes duration, with minimum interval of 24 hours, for a period of 8 weeks. Each session will consist of three parts: aerobic training, strength training and respiratory physiotherapy. The aerobic training will be held for 35 minutes (10 min of warm up, 20 min on target load and 5 min of slowdown) with initial intensity of 60% of the maximum load obtained in the maximal cardiopulmonary exercise testing or in incremental shuttle walk test (ISWT). The intensity will be gradually increased up to 80%, so that fatigue or dyspnea values are kept between 4 and 6, according to the modified Borg scale.
  Interventions: Other: Intervention Group
- Control Group (Active Comparator): The control group will be subjected to supervised respiratory physiotherapy and stretching exercises twice a week, each session with duration of 60 minutes, with minimum interval of 24 hours, for a period of 8 weeks. The oral high-frequency oscillation device (Flutter®) will be used for 10 minutes, 5 minutes in each lateral decubitus, followed by the stretching of upper and lower limbs for 40 minutes. All exercises will be active, performed in sitting and lying positions without increasing the heart rate. The remaining 10 minutes will be used to discuss doubts about the disease and the use of the booklet.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Intervention Group — Aerobic training
  Other Names: Pulmonary Rehabilitation
  Arms: Intervention Group
Other: Control Group — Chest physiotherapy: Flutter and muscle stretching
  Other Names: Chest Physiotherapy
  Arms: Control Group

SUMMARY:
Asthma is one of the main chronic diseases in childhood and it is characterized by the inflammation of airways. Individuals with chronic lung disease are more susceptible to present reduction in exercise tolerance due to pulmonary limitations. The pulmonary rehabilitation may improve the physical capacity in asthmatic patients, as observed in other chronic lung diseases.

DETAILED DESCRIPTION:
The asthmatic patient's clinical changes may impair their functional capacity and exercise tolerance. Thus, the treatment of these individuals should be extended to pulmonary rehabilitation. Randomized clinical trials have shown interesting results, whether in cardiopulmonary conditions, quality of life or in the number of crises, after applying pulmonary rehabilitation program in asthmatic children and adolescents. In a systematic review on physical training with asthmatic children and adolescents the authors concluded that physical activity should be recommended to this population, although some issues have not yet been clarified due to limitations in the clinical trial. The control of the disease has not been evaluated by specific questionnaires in any study. The assessment of inflammatory markers was rarely addressed and the same occurred in the quality of life after physical training. In addition, it is possible to question the intensity and frequency of training, factors that can significantly contribute to the intervention results. All these information let us know that is necessary a randomized control trial to answer questions about physical characteristics, quality of life, inflammatory markers, and muscles strength.

ELIGIBILITY:
Inclusion Criteria:

* between six and 18 years old
* asthma-diagnosed patients
* under medical treatment and disease control

Exclusion Criteria:

* fail to carry out the protocol evaluations
* interrupt the medical care and/or drug-based treatment
* acute lung infection or other chronic lung diseases
* other comorbidities (neuropathies, heart disease)
* missing in more than 20% the rehabilitation protocol

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Physical capacity as measure by distance walked of shuttle walk test and oxygen consumption (VO2) | Physiscal capacity will be measured at the beginning and at the end of the protocol (after 8 weeks)
  Modified shuttle test was conducted

SECONDARY OUTCOMES:
Muscle strength as measure by electromyography (EMG) | Muscles strenght will be measured at the begening and at the end of the protocol (after 8 weeks).
  1 maximal repetition was performed
Muscle endurance as measure by electromyography (EMG) | Muscles endurance will be measured at the begening and at the end of the protocol (after 8 weeks).
Quality of life measured by Pediatric questionnaire | Quesitionnaire will be measured at the begening and at the end of the protocol (after 8 weeks).
Inflammatory markers as measure by interleukines | Inflamatory markers will be measured at the begening and at the end of the protocol (after 8 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Dirceu Solé, PhD, Study Chair — Unifesp, Federal University of Sao Paulo
Locations (1):
- Fernanda C Lanza, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Silva EP, Soares BA, Reimberg MM, Ritti-Dias R, Nascimento KS, Anjos FS, Wandalsen GF, Sole D, Dal Corso S, Lanza FC. Heart rate recovery in asthmastic children and adolescents after clinical field test. BMC Pulm Med. 2021 Feb 19;21(1):61. doi: 10.1186/s12890-020-01355-9. PMID 33607978
- [Derived] Reimberg MM, Castro RA, Selman JP, Meneses AS, Politti F, Mallozi MC, Wandalsen GF, Sole D, De Angelis K, Dal Corso S, Lanza FC. Effects of a pulmonary rehabilitation program on physical capacity, peripheral muscle function and inflammatory markers in asthmatic children and adolescents: study protocol for a randomized controlled trial. Trials. 2015 Aug 13;16:346. doi: 10.1186/s13063-015-0876-x. PMID 26268930